CLINICAL TRIAL: NCT02977767
Title: Evaluation of the Effect of Conversational Hypnosis When Changing Tracheal Cannula in Adult Patients: a Pilot Study
Brief Title: Evaluation of the Effect of Conversational Hypnosis When Changing Tracheal Cannula in Adult Patients
Acronym: HYPNO-TRACH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants do not accept hypnosis.
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/CHU/02
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Tracheotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversational hypnosis (Experimental): Use of conversational hypnosis during the tracheal cannula replacement
  Interventions: Procedure: Conversational hypnosis

INTERVENTIONS:
Procedure: Conversational hypnosis — Conversational hypnosis starts since the enter of the nurse in patient's room and last since the nurse leaves the room. Change of canula is performed under conversational hypnosis.

SUMMARY:
Tracheotomy is requested when upper aero-digestive tracts are obstructed. This obstruction can have a tumour, infectious, inflammatory, traumatic or nervous origin. Most tracheotomy surgeries are performed for tumour-induced obstruction. Tracheotomy allows the setting of a respiratory flux thanks to a cannula and excludes the upper airways. The cannula is washed every day from once to several times depending on the patient's secretions production and it is usually replaced every week. The second replacement takes place about 10 days after surgery. Patient education takes place at every replacement in order to empower him/her and in consequence to increase living comfort. This empowerment is achieved at the 4th or 5th replacement, at best. Because of the risks and complications related to tracheotomy and because of the concerned vital function, the cannula replacement leads to anxiety especially during the first replacements. Usual patient's anxiety management consists in reassuring the patient during the replacement. In other situations, patients' anxiety management would be drugs, however due to sedative and anxiolytic drugs' adverse events and to the need to maintain optimal breathing, they are not used in first intention. Our choice is to use conversational hypnosis during cannula replacement as it has already demonstrated interesting effects in pain and anxiety. Conversational hypnosis does not present an induction phase like in so-called hypnosis, it aims at leading the patient to perceive his/her world differently with only a slight consciousness alteration.

DETAILED DESCRIPTION:
Once the informed consent form is signed and when the cannula replacement has to be performed, conversational hypnosis session will start right from the patient's room entrance and end when the nurse will come out. The care will consist in aspiration, cleaning and finally replacement of the cannula. Adverse events are expected to be related to the cannula replacement itself: patients will be followed-up during a maximum of 7 days with one follow-up visit which will take place 2 hours after cannula replacement and a second one which can take place from the day after the replacement up to just before the following replacement.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalised in the Ear, Nose, Throat - specialties surgery department
* aged of 18 years old and more
* having a tracheotomy following an upper aero-digestive tracts obstruction
* presenting a tracheal cannula which can be replaced by paramedical staff
* able to communicate to give their consent
* member or beneficiary of a social security assurance
* having given a signed informed consent form

Exclusion Criteria:

* patients presenting a hearing loss (preventing from hearing properly the words pronounced during conversational hypnosis)
* who do not understand French
* who are under curators/guardianship
* presenting dementia
* autonomous in their cannula replacement
* having already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Time to change the tracheal cannula using conversational hypnosis | On the patient's scope, time measured from the moment the nurse says "now we start" according to the conversational hypnosis protocol to the time the new cannula is fixed around the patient's neck, assessed up to 1 hour (3600 seconds).
  Once the written informed consent form is obtained, the tracheal cannula change to perform in the frame of the study can be performed. As the patient will be scoped, the time to change the cannula will be monitored: the nurse will use an indicator on the scope to mark the start of the cannula change (when the sentence "now we start" is pronounced according to the conversational hypnosis protocol) and an indicator is placed on the scope when the new cannula is fixed around the patient's neck. The time between the two indicators will be reported in the Case Report Form in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Daw-Horng WU, MD, Principal Investigator — CHU La Réunion

IPD SHARING:
Plan to Share IPD: No